CLINICAL TRIAL: NCT02755558
Title: Effects of Energy Density and Portion Size of Milk in Preschool Children
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Penn State University (Other)
Collaborators: National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK) (NIH)
Responsible Party: Principal Investigator, Barbara J. Rolls, Professor of Nutritional Sciences, Penn State University
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Basic Science
Other Study IDs: ChildFood301; R01DK082580 (NIH); 2011-67001-30117 (Other Grant/Funding Number: The Pennsylvania State University)
Record Dates: First submitted 2016-04-22; First posted 2016-04-29 (Estimated); Last update posted 2017-03-21 (Actual); Status verified 2017-03

CONDITIONS: Feeding Behaviors
MeSH Terms: conditions — Feeding Behavior

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (4):
- Low energy density, small portion (Experimental): Low milk energy density and small portion size
  Interventions: Behavioral: Low energy density; Behavioral: Small portion
- Low energy density, large portion (Experimental): Low milk energy density and large portion size
  Interventions: Behavioral: Low energy density; Behavioral: Large portion
- High energy density, small portion (Experimental): High milk energy density and small portion size
  Interventions: Behavioral: High energy density; Behavioral: Small portion
- High energy density, large portion (Experimental): High milk energy density and large portion size
  Interventions: Behavioral: High energy density; Behavioral: Large portion

INTERVENTIONS:
Behavioral: Low energy density — Low energy density milk served
  Arms: Low energy density, large portion; Low energy density, small portion
Behavioral: High energy density — High energy density milk served
  Arms: High energy density, large portion; High energy density, small portion
Behavioral: Small portion — Small portion of milk served
  Arms: High energy density, small portion; Low energy density, small portion
Behavioral: Large portion — Large portion of milk served
  Arms: High energy density, large portion; Low energy density, large portion

SUMMARY:
In this study, the investigators varied both the energy density and portion size of milk served with a meal commonly consumed by preschool children. The milk used in this study is commercially available and reflects typical variations in energy density. The primary aim of the study is to investigate the independent and combined effects of milk energy density and portion size on preschool children's intake of the milk and the simultaneously served meal. The effect of milk energy density and portion size on children's total energy intake at the meal will also be evaluated.

ELIGIBILITY:
Inclusion Criteria:

* Children must be enrolled in participating childcare centers

Exclusion Criteria:

* Allergy or intolerance to any of the foods or beverages served

Ages: 3 Years to 6 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 143 (Actual)
Dates: Start 2014-09; Primary Completion 2015-05 (Actual); Study Completion 2015-05 (Actual)

PRIMARY OUTCOMES:
Difference between experimental conditions for milk, food, and total intake by weight | once a week for 4 weeks
  Difference between experimental conditions in milk intake (weight in grams), food intake (weight in grams), total meal intake (weight in grams)
Difference between experiential conditions for milk, food, and total intake by energy | once a week for 4 weeks
  Difference between experimental conditions for milk intake (energy in kcal), food intake (energy in kcal), and total meal energy intake (energy in kcal)

SECONDARY OUTCOMES:
Meal energy density | once a week for 4 weeks
  Meal energy density (energy density in kcal/g)

CONTACTS AND LOCATIONS:
Overall Officials: Barbara J Rolls, Principal Investigator — The Pennsylvania State University
Locations (1):
- The Pennsylvania State University, Laboratory for the Study of Human Ingestive Behavior, University Park, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: Undecided